CLINICAL TRIAL: NCT04856917
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Participants With Acne Vulgaris
Brief Title: A Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Participants With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB019-209
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-05

CONDITIONS: Acne Vulgaris
Keywords: LI-36 Receptor; Interleukin 36; Imsidolimab
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Imsidolimab 400/200 mg (Experimental): Participants received imsidolimab 400 milligrams (mg) by subcutaneous (SC) injection on Day 1, followed by 200 mg on Days 29 and 57.
  Interventions: Drug: Imsidolimab
- Imsidolimab 200/100 mg (Experimental): Participants received imsidolimab 200 mg by SC injection on Day 1, followed by 100 mg on Days 29 and 57.
  Interventions: Drug: Imsidolimab
- Placebo (Placebo Comparator): Participants received imsidolimab matching placebo by SC injection on Days 1, 29, and 57.
  Interventions: Biological: Placebo

INTERVENTIONS:
Drug: Imsidolimab — Humanized Monoclonal Antibody
  Other Names: ANB019
  Arms: Imsidolimab 200/100 mg; Imsidolimab 400/200 mg
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy and Safety of Imsidolimab in Participants with Acne Vulgaris

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of imsidolimab in adolescent and adult participants with acne vulgaris (AV). This study also will characterize the pharmacokinetic (PK) profile of imsidolimab and explore the immune response to imsidolimab in participants with AV.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of moderate to severe facial AV
* Facial IGA) score of 3 (moderate) or 4 (severe)
* At least 20 and no more than 100 inflammatory lesions on the face
* No more than 100 non-inflammatory lesions on the face.
* No more than 5 nodules (≥5 millimeter [mm]) on the face

Key Exclusion Criteria:

* A participant with acne fulminans or conglobate or secondary acne will be excluded.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - Site 10-114, Hot Springs, Arkansas
  - Site 10-111, Fountain Valley, California
  - Site 10-106, Sherman Oaks, California
  - Site 10-113, Sweetwater, Florida
  - Site 10-108, Tampa, Florida
  - Site 10-107, Tampa, Florida
  - Site 10-109, New Orleans, Louisiana
  - Site 10-112, New Orleans, Louisiana
  - Site 10-104, Detroit, Michigan
  - Site 10-110, Portsmouth, New Hampshire
  - Site 10-105, Murfreesboro, Tennessee
  - Site 10-103, Austin, Texas
  - Site 10-102, College Station, Texas
  - Site 10-101, San Antonio, Texas
- Site 10-115, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Started | 42 | 40 | 41
Safety Analysis Set (The Safety Analysis Set included all randomized participants who received at least 1 dose of imsidolimab or placebo.) | 41 | 39 | 41
Completed | 34 | 34 | 37
Not Completed | 8 | 6 | 4
Not completed — Withdrawal by Subject | 4 | 3 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Used of Prohibited Medication or Treatment | 0 | 1 | 2
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized participants.
Groups:
- Imsidolimab 400/200 mg: Participants received imsidolimab 400 mg by SC injection on Day 1, followed by 200 mg on Days 29 and 57.
- Total: Total of all reporting groups
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo | Total
Number analyzed (Participants) | 42 | 40 | 41 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.3 (5.58) | 20.7 (7.39) | 21.0 (7.62) | 20.3 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 26 | 80
  Male | 18 | 10 | 15 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 13 | 11 | 41
  Not Hispanic or Latino | 25 | 27 | 30 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 9 | 22
  White | 34 | 28 | 31 | 93
  More than one race | 2 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Facial inflammatory Lesion Count [Mean (Standard Deviation); unit: lesions] — The number of facial inflammatory lesions (pustules, papules, and nodular lesions) on the forehead, left and right cheeks, nose, and chin were counted. Baseline was defined as the last available measurement taken prior to the first dose of study treatment.
  lesions | 29.5 (8.12) | 29.0 (12.34) | 26.9 (7.11) | 28.5 (9.42)
Facial Investigator's Global Assessment (IGA) score [Mean (Standard Deviation); unit: units on a scale] — It is a 5-point morphological assessment ranging from 0 (clear) to 4 (severe).
  Clear (0): clear skin with no inflammatory or non-inflammatory lesions
  Almost Clear (1): A few scattered comedones and a few small papules
  Mild (2): Easily recognizable; less than half the surface is involved. some comedones and some papules and pustules
  Moderate (3): More than half of the surface is involved. Many comedones, papules, and pustules. One nodule may be present
  Severe (4): Entire surface is involved. Covered with comedones, numerous papules and pustules. Few nodules may be present.
  units on a scale | 3.1 (0.35) | 3.1 (0.27) | 3.1 (0.33) | 3.1 (0.32)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Facial Inflammatory Lesion Counts at Week 12
Description: The number of facial inflammatory lesions (pustules, papules, and nodular lesions) on the forehead, left and right cheeks, nose, and chin were counted. Baseline was defined as the last available measurement taken prior to the first dose of study treatment.
Time Frame: Baseline, Week 12
Population: Participants in ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 34 | 35 | 36
lesions | -6.8 (13.63) | -7.4 (16.38) | -9.6 (10.66)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Least square (LS) Mean, SE, 90% CI, & p-value was based on a linear repeated measures model (LRMM) which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline facial inflammatory lesion count as continuous covariate; Test type: Superiority; p = 0.3757, LRMM; LS Mean Difference = 2.9, 90% CI 2-sided [-2.47 to 8.19], Standard Error of Mean 3.21
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; LS Mean, SE, 90% CI, & p-value was based on a LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline facial inflammatory lesion count as continuous covariate; Test type: Superiority; p = 0.6183, LRMM; LS Mean Difference = 1.6, 90% CI 2-sided [-3.73 to 6.95], Standard Error of Mean 3.22

2. Secondary Outcome: Change From Baseline in Facial Inflammatory Lesion Counts at Weeks 2, 4, 8, and 20
Description: as for outcome 1
Time Frame: Baseline, Weeks 2, 4, 8, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Imsidolimab 400/200 mg: Participants received imsidolimab 400mg by SC injection on Day 1, followed by 200 mg on Days 29 and 57.
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
lesions
  Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Change at Week 2 | -1.9 (7.87) | -0.5 (7.30) | -3.8 (7.04)
  Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Change at Week 4 | -0.3 (15.21) | -4.4 (9.87) | -8.0 (9.64)
  Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Change at Week 8 | -5.5 (10.75) | -6.2 (12.43) | -7.8 (12.40)
  Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Change at Week 20 | -8.7 (11.42) | -12.0 (16.58) | -11.7 (9.00)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.2490, LRMM — LS Mean, SE, 90% CI, & p-value was based on a LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline facial inflammatory lesion count as continuous covariate; LS Mean Difference = 2.0, 90% CI 2-sided [-0.85 to 4.80], Standard Error of Mean 1.70
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.0708, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 3.1, 90% CI 2-sided [0.28 to 5.99], Standard Error of Mean 1.72
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0040, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 7.9, 90% CI 2-sided [3.44 to 12.34], Standard Error of Mean 2.68
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.2060, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 3.4, 90% CI 2-sided [-1.05 to 7.94], Standard Error of Mean 2.71
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.4341, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 2.1, 90% CI 2-sided [-2.33 to 6.51], Standard Error of Mean 2.66
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.7307, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.9, 90% CI 2-sided [-3.59 to 5.48], Standard Error of Mean 2.73
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.3261, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 2.9, 90% CI 2-sided [-1.97 to 7.77], Standard Error of Mean 2.93
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.8221, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.7, 90% CI 2-sided [-5.56 to 4.23], Standard Error of Mean 2.95

3. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory Lesion Counts at Weeks 2, 4, 8, 12, and 20
Description: as for outcome 1
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
percent change
  Percent Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Percent Change at Week 2 | -6.6 (27.87) | -1.9 (27.37) | -13.6 (25.76)
  Percent Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Percent Change at Week 4 | -2.9 (44.00) | -14.1 (31.98) | -29.3 (33.39)
  Percent Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Percent Change at Week 8 | -21.50 (33.89) | -19.6 (39.15) | -28.4 (42.87)
  Percent Change at Week 12: number analyzed (Participants) | 34 | 35 | 36
  Percent Change at Week 12 | -26.8 (42.68) | -20.5 (53.96) | -37.6 (40.73)
  Percent Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Percent Change at Week 20 | -34.3 (37.50) | -36.4 (48.53) | -46.9 (32.95)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.3008, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 6.4, 90% CI 2-sided [-3.84 to 16.73], Standard Error of Mean 6.20
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.0878, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 10.8, 90% CI 2-sided [0.40 to 21.19], Standard Error of Mean 6.27
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0020, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 26.6, 90% CI 2-sided [12.64 to 40.57], Standard Error of Mean 8.42
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.1029, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 14.0, 90% CI 2-sided [-0.12 to 28.09], Standard Error of Mean 8.50
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.5427, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 5.4, 90% CI 2-sided [-9.25 to 20.02], Standard Error of Mean 8.82
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.5833, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 5.0, 90% CI 2-sided [-10.05 to 20.02], Standard Error of Mean 9.06
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.3293, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 10.8, 90% CI 2-sided [-7.46 to 28.99], Standard Error of Mean 10.98
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.1900, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 14.5, 90% CI 2-sided [-3.74 to 32.74], Standard Error of Mean 10.99
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.2168, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 11.7, 90% CI 2-sided [-3.91 to 27.23], Standard Error of Mean 9.38
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.4089, LRMM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 7.8, 90% CI 2-sided [-7.82 to 23.45], Standard Error of Mean 9.42

4. Secondary Outcome: Change From Baseline in Facial Non-inflammatory Lesion Counts at Weeks 2, 4, 8, 12, and 20
Description: The number of facial non-inflammatory lesions (open and closed comedones) on the forehead, left and right cheeks, and chin was counted. Baseline was defined as the last available measurement taken prior to the first dose of study treatment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
lesions
  Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Change at Week 2 | -2.2 (11.28) | -0.9 (9.95) | -3.2 (14.07)
  Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Change at Week 4 | -4.7 (11.87) | -4.3 (10.15) | -6.4 (14.98)
  Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Change at Week 8 | -6.5 (21.57) | -2.2 (16.65) | -8.1 (15.30)
  Change at Week 12: number analyzed (Participants) | 34 | 35 | 36
  Change at Week 12 | -6.6 (20.18) | -4.5 (17.89) | -9.4 (16.96)
  Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Change at Week 20 | -9.9 (15.31) | -4.0 (20.90) | -11.0 (15.01)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.4229, LRMM — LS Mean, SE, 90% CI, & p-value was based on LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs 4) as categorical covariates & baseline facial non-inflammatory lesion count as continuous covariate; LS Mean Difference = 2.0, 90% CI 2-sided [-2.16 to 6.24], Standard Error of Mean 2.53
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.6027, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 1.3, 90% CI 2-sided [-2.91 to 5.59], Standard Error of Mean 2.56
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.2655, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 2.8, 90% CI 2-sided [-1.35 to 6.95], Standard Error of Mean 2.50
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.6229, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 1.2, 90% CI 2-sided [-2.95 to 5.44], Standard Error of Mean 2.53
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.4091, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 3.1, 90% CI 2-sided [-3.10 to 9.30], Standard Error of Mean 3.74
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.1274, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 5.9, 90% CI 2-sided [-0.47 to 12.25], Standard Error of Mean 3.83
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.2075, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 4.8, 90% CI 2-sided [-1.47 to 11.01], Standard Error of Mean 3.76
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.2484, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 4.4, 90% CI 2-sided [-1.88 to 10.64], Standard Error of Mean 3.77
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.3399, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 3.5, 90% CI 2-sided [-2.53 to 9.45], Standard Error of Mean 3.61
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.0545, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 7.0, 90% CI 2-sided [1.03 to 13.05], Standard Error of Mean 3.62

5. Secondary Outcome: Percent Change From Baseline in Facial Non-Inflammatory Lesion Counts at Weeks 2, 4, 8, 12, and 20
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
percent change
  Percent Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Percent Change at Week 2 | -1.0 (37.86) | 1.0 (49.80) | 1.1 (67.11)
  Percent Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Percent Change at Week 4 | -6.8 (37.46) | -8.7 (45.48) | -12.7 (45.88)
  Percent Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Percent Change at Week 8 | -7.7 (84.17) | 11.4 (117.96) | -18.1 (32.73)
  Percent Change at Week 12: number analyzed (Participants) | 34 | 35 | 36
  Percent Change at Week 12 | -2.4 (68.07) | 8.8 (114.44) | -22.1 (40.26)
  Percent Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Percent Change at Week 20 | -21.1 (46.59) | -0.9 (95.05) | -31.4 (50.91)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.9679, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.5, 90% CI 2-sided [-19.86 to 18.91], Standard Error of Mean 11.69
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.9152, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -1.3, 90% CI 2-sided [-20.87 to 18.35], Standard Error of Mean 11.83
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.4490, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 7.3, 90% CI 2-sided [-8.67 to 23.32], Standard Error of Mean 9.64
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.7246, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 3.4, 90% CI 2-sided [-12.72 to 19.60], Standard Error of Mean 9.74
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.4655, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 13.8, 90% CI 2-sided [-17.49 to 45.14], Standard Error of Mean 18.88
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.1178, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 30.5, 90% CI 2-sided [-1.59 to 62.54], Standard Error of Mean 19.33
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.1938, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 23.1, 90% CI 2-sided [-6.22 to 52.52], Standard Error of Mean 17.71
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.0991, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 29.7, 90% CI 2-sided [0.08 to 59.29], Standard Error of Mean 17.85
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.3337, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 15.0, 90% CI 2-sided [-10.62 to 40.59], Standard Error of Mean 15.44
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.0465, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 31.2, 90% CI 2-sided [5.50 to 56.87], Standard Error of Mean 15.48

6. Secondary Outcome: Change From Baseline in Total Facial Lesion (Inflammatory and Non-inflammatory Lesions) Counts at Weeks 2, 4, 8, 12, and 20
Description: The number of facial inflammatory (pustules, papules, and nodular lesions) and non-inflammatory (open and closed comedones) lesions on the forehead, left and right cheeks, nose, and chin were counted. Baseline was defined as the last available measurement taken prior to the first dose of study treatment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
lesions
  Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Change at Week 2 | -4.1 (15.03) | -1.3 (11.95) | -7.0 (12.36)
  Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Change at Week 4 | -5.0 (21.03) | -8.7 (16.32) | -14.4 (15.22)
  Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Change at Week 8 | -12.0 (28.0) | -8.4 (23.85) | -15.9 (19.50)
  Change at Week 12: number analyzed (Participants) | 34 | 35 | 36
  Change at Week 12 | -13.4 (26.82) | -11.9 (29.06) | -19.0 (21.24)
  Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Change at Week 20 | -18.6 (22.01) | -16.0 (31.82) | -22.7 (18.65)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.2150, LRMM — LS Mean, SE, 90% CI, & p-value was based on a LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline total facial lesion count as continuous covariate; LS Mean Difference = 3.7, 90% CI 2-sided [-1.21 to 8.56], Standard Error of Mean 2.95
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.0864, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 5.1, 90% CI 2-sided [0.21 to 10.05], Standard Error of Mean 2.97
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0084, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 10.4, 90% CI 2-sided [3.97 to 16.85], Standard Error of Mean 3.88
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.1600, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 5.5, 90% CI 2-sided [-0.95 to 12.01], Standard Error of Mean 3.91
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.3671, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 4.7, 90% CI 2-sided [-3.94 to 13.41], Standard Error of Mean 5.23
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.1587, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 7.6, 90% CI 2-sided [-1.28 to 16.46], Standard Error of Mean 5.35
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.1932, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 7.6, 90% CI 2-sided [-2.03 to 17.21], Standard Error of Mean 5.80
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.2518, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 6.7, 90% CI 2-sided [-2.95 to 16.37], Standard Error of Mean 5.82
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.2320, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 6.7, 90% CI 2-sided [-2.53 to 15.83], Standard Error of Mean 5.53
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.2014, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 7.1, 90% CI 2-sided [-2.08 to 16.35], Standard Error of Mean 5.55

7. Secondary Outcome: Percent Change From Baseline in Total Facial Lesion (Inflammatory and Non-inflammatory Lesions) Counts at Weeks 2, 4, 8, 12, and 20
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
percent change
  Percent Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Percent Change at Week 2 | -6.9 (21.26) | -1.9 (21.62) | -10.7 (22.27)
  Percent Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Percent Change at Week 4 | -7.7 (29.10) | -13.5 (22.61) | -23.2 (23.87)
  Percent Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Percent Change at Week 8 | -18.9 (40.88) | -12.7 (31.36) | -24.0 (27.82)
  Percent Change at Week 12: number analyzed (Participants) | 34 | 35 | 36
  Percent Change at Week 12 | -18.9 (39.18) | -15.4 (44.85) | -31.2 (31.88)
  Percent Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Percent Change at Week 20 | -28.6 (33.69) | -23.0 (56.30) | -38.7 (30.00)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.4361, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 3.9, 90% CI 2-sided [-4.34 to 12.06], Standard Error of Mean 4.94
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.1018, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 8.2, 90% CI 2-sided [-0.04 to 16.48], Standard Error of Mean 4.98
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0059, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 16.3, 90% CI 2-sided [6.66 to 25.88], Standard Error of Mean 5.79
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0913, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 9.9, 90% CI 2-sided [0.26 to 19.59], Standard Error of Mean 5.83
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.4921, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 5.3, 90% CI 2-sided [-7.47 to 18.09], Standard Error of Mean 7.70
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.1607, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 11.1, 90% CI 2-sided [-1.95 to 24.24], Standard Error of Mean 7.89
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.1244, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 14.2, 90% CI 2-sided [-1.02 to 29.48], Standard Error of Mean 9.19
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.1004, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 15.2, 90% CI 2-sided [-0.02 to 30.51], Standard Error of Mean 9.20
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.2015, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 12.4, 90% CI 2-sided [-3.61 to 28.39], Standard Error of Mean 9.64
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.1057, LRMM — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 15.8, 90% CI 2-sided [-0.27 to 31.81], Standard Error of Mean 9.66

8. Secondary Outcome: Change From Baseline in Facial Investigator's Global Assessment (IGA) at Weeks 2, 4, 8, 12, and 20
Description: The Facial IGA was a global assessment that was used to assess the current state of acne vulgaris (AV) on the face at each visit. It is a 5-point morphological assessment ranging from 0 (clear) to 4 (severe).
  Clear (0): clear skin with no inflammatory or non-inflammatory lesions
  Almost Clear (1): A few scattered comedowns and a few small papules
  Mild (2): Easily recognizable; less than half the surface is involved. some comedowns and some papules and pustules
  Moderate (3): More than half of the surface is involved. Many comedowns, papules, and pustules. One nodule may be present
  Severe (4): Entire surface is involved. Covered with comedowns, numerous papules and pustules. Few nodules may be present.
  The Facial IGA was an overall global evaluation that was performed at an arm's length distance from the participant and must be performed before the acne lesion count.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
units on a scale
  Change at Week 2: number analyzed (Participants) | 40 | 38 | 38
  Change at Week 2 | -0.2 (0.46) | -0.0 (0.16) | -0.2 (0.43)
  Change at Week 4: number analyzed (Participants) | 38 | 37 | 39
  Change at Week 4 | -0.2 (0.49) | -0.1 (0.42) | -0.5 (0.60)
  Change at Week 8: number analyzed (Participants) | 40 | 35 | 38
  Change at Week 8 | -0.4 (0.62) | -0.3 (0.53) | -0.6 (0.60)
  Change at Week 12: number analyzed (Participants) | 34 | 35 | 36
  Change at Week 12 | -0.6 (0.78) | -0.3 (0.54) | -0.8 (0.83)
  Change at Week 20: number analyzed (Participants) | 35 | 35 | 37
  Change at Week 20 | -0.7 (0.91) | -0.7 (0.80) | -0.9 (0.71)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.5157, LRMM — LS Mean, SE, 90% CI, & p-value was based on a LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline facial IGA as continuous covariate; LS Mean Difference = 0.1, 90% CI 2-sided [-0.08 to 0.19], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.0178, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.2, 90% CI 2-sided [0.06 to 0.34], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0132, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.3, 90% CI 2-sided [0.10 to 0.48], Standard Deviation 0.12
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0034, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.3, 90% CI 2-sided [0.16 to 0.54], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.0510, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.3, 90% CI 2-sided [0.04 to 0.47], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.0608, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.3, 90% CI 2-sided [0.03 to 0.47], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.2702, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.2, 90% CI 2-sided [-0.10 to 0.48], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.0249, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.4, 90% CI 2-sided [0.11 to 0.69], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.1853, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.2, 90% CI 2-sided [-0.06 to 0.55], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.2974, LRMM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.2, 90% CI 2-sided [-0.11 to 0.50], Standard Error of Mean 0.18

9. Secondary Outcome: Percentage of Participants Achieving a Facial IGA of Clear (0) or Almost Clear (1) With at Least a 2-grade Decrease From Baseline at Weeks 2, 4, 8, 12, and 20
Description: The Facial IGA was a global assessment that was used to assess the current state of AV on the face at each visit. It is a 5-point morphological assessment ranging from 0 (clear) to 4 (severe).
  Clear (0): clear skin with no inflammatory or non-inflammatory lesions
  Almost Clear (1): A few scattered comedowns and a few small papules
  Mild (2): Easily recognizable; less than half the surface is involved. some comedowns and some papules and pustules
  Moderate (3): More than half of the surface is involved. Many comedowns, papules, and pustules. One nodule may be present
  Severe (4): Entire surface is involved. Covered with comedowns, numerous papules and pustules. Few nodules may be present.
  The Facial IGA was an overall global evaluation that was performed at an arm's length distance from the participant and must be performed before the acne lesion count.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
percentage of participants
  Week 2: number analyzed (Participants) | 40 | 38 | 38
  Week 2 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 38 | 37 | 39
  Week 4 | 0 | 0 | 2.6
  Week 8: number analyzed (Participants) | 40 | 35 | 38
  Week 8 | 2.5 | 0 | 2.6
  Week 12: number analyzed (Participants) | 34 | 35 | 36
  Week 12 | 11.8 | 0 | 13.9
  Week 20: number analyzed (Participants) | 35 | 35 | 37
  Week 20 | 14.3 | 8.6 | 18.9
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.3390, Cochran-Mantel-Haenszel — P-value for the adjusted risk difference between imsidolimab and placebo was obtained from generalized Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA score at baseline; Risk Difference (RD) = -2.50, 90% CI 2-sided [-6.62 to 1.63]
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.3243, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = -2.60, 90% CI 2-sided [-6.79 to 1.59]
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = 0.00, 90% CI 2-sided [-5.91 to 5.91]
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.3320, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = -2.66, 90% CI 2-sided [-6.96 to 1.63]
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.7595, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = -2.45, 90% CI 2-sided [-15.50 to 10.59]
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.0209, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = -14.11, 90% CI 2-sided [-23.66 to -4.57]
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.6094, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = -4.56, 90% CI 2-sided [-18.99 to 9.87]
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.2076, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Risk Difference (RD) = -10.28, 90% CI 2-sided [-23.34 to 2.78]

10. Secondary Outcome: Percentage of Participants in Each Response Category for the Patient Global Impression of Severity (PGI-S) at Weeks 2, 4, 8, 12, and 20
Description: PGI- S was a single-item question, which asks the participant to rate the current severity of AV. The response options were:
  Clear Skin (1)
  Mild (2)
  Moderate (3)
  Severe (4)
  Higher score indicated more severity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
percentage of participants
  Week 2: Clear Skin: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Clear Skin | 0 | 0 | 0
  Week 2: Mild: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Mild | 25.0 | 23.7 | 21.1
  Week 2: Moderate: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Moderate | 55.0 | 63.2 | 50.0
  Week 2: Severe: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Severe | 20.0 | 13.2 | 28.9
  Week 4: Clear Skin: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Clear Skin | 0 | 0 | 0
  Week 4: Mild: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Mild | 26.3 | 21.6 | 33.3
  Week 4: Moderate: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Moderate | 63.2 | 70.3 | 48.7
  Week 4: Severe: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Severe | 10.5 | 8.1 | 17.9
  Week 8: Clear Skin: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Clear Skin | 2.5 | 0 | 0
  Week 8: Mild: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Mild | 27.5 | 48.6 | 44.7
  Week 8: Moderate: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Moderate | 60.0 | 45.7 | 47.4
  Week 8: Severe: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Severe | 10.0 | 5.7 | 7.9
  Week 12: Clear Skin: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Clear Skin | 5.9 | 0 | 0
  Week 12: Mild: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Mild | 41.2 | 42.9 | 50.0
  Week 12: Moderate: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Moderate | 44.1 | 51.4 | 47.2
  Week 12: Severe: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Severe | 8.8 | 5.7 | 2.8
  Week 20: Clear Skin: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Clear Skin | 2.9 | 2.9 | 2.6
  Week 20: Mild: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Mild | 54.3 | 57.1 | 63.2
  Week 20: Moderate: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Moderate | 34.3 | 34.3 | 28.9
  Week 20: Severe: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Severe | 8.6 | 5.7 | 5.3
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.4482, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = 0.10, 90% CI 2-sided [-0.10 to 0.29] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.4529, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = 0.14, 90% CI 2-sided [-0.05 to 0.33] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.9320, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.01, 90% CI 2-sided [-0.20 to 0.18] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.3151, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.03, 90% CI 2-sided [-0.22 to 0.16] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.2908, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.14, 90% CI 2-sided [-0.32 to 0.06] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.7277, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.15 to 0.24] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.8463, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.03, 90% CI 2-sided [-0.23 to 0.17] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.5281, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.08, 90% CI 2-sided [-0.28 to 0.11] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.5747, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.09, 90% CI 2-sided [-0.28 to 0.11] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.5081, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.05, 90% CI 2-sided [-0.24 to 0.14] — Somers'D statistic and tanh^(-1) transformed 90% CI

11. Secondary Outcome: Percentage of Participants in Each Response Category for the Patient Global Impression of Change (PGI-C) at Weeks 2, 4, 8, 12, and 20
Description: PGI-C was a single-item, self-administered questionnaire, which asked the participant to rate the change in their symptom severity. Scores ranged from 1 (Very much better) to 7 (Very much worse).
  Very much better (1)
  Much better (2)
  A little better (3)
  No change (4)
  A little worse (5)
  Much worse (6)
  Very much worse (7)
  Higher score indicated more severity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 39
percentage of participants
  Week 2: Very much better: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Very much better | 0 | 0 | 0
  Week 2: Much better: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Much better | 5.0 | 2.6 | 2.6
  Week 2: A little better: number analyzed (Participants) | 40 | 38 | 38
  Week 2: A little better | 55.0 | 50.0 | 52.6
  Week 2: No change: number analyzed (Participants) | 40 | 38 | 38
  Week 2: No change | 20.0 | 18.4 | 34.2
  Week 2: A little worse: number analyzed (Participants) | 40 | 38 | 38
  Week 2: A little worse | 15.0 | 18.4 | 10.5
  Week 2: Much worse: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Much worse | 5.0 | 10.5 | 0
  Week 2: Very much worse: number analyzed (Participants) | 40 | 38 | 38
  Week 2: Very much worse | 0 | 0 | 0
  Week 4: Very much better: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Very much better | 0 | 2.7 | 0
  Week 4: Much better: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Much better | 7.9 | 13.5 | 15.4
  Week 4: A little better: number analyzed (Participants) | 38 | 37 | 39
  Week 4: A little better | 47.4 | 37.8 | 56.4
  Week 4: No change: number analyzed (Participants) | 38 | 37 | 39
  Week 4: No change | 26.3 | 18.9 | 15.4
  Week 4: A little worse: number analyzed (Participants) | 38 | 37 | 39
  Week 4: A little worse | 13.2 | 16.2 | 12.8
  Week 4: Much worse: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Much worse | 2.6 | 8.1 | 0
  Week 4: Very much worse: number analyzed (Participants) | 38 | 37 | 39
  Week 4: Very much worse | 2.6 | 2.7 | 0
  Week 8: Very much better: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Very much better | 5.0 | 2.9 | 2.6
  Week 8: Much better: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Much better | 17.5 | 14.3 | 31.6
  Week 8: A little better: number analyzed (Participants) | 40 | 35 | 38
  Week 8: A little better | 47.5 | 40.0 | 50.0
  Week 8: No change: number analyzed (Participants) | 40 | 35 | 38
  Week 8: No change | 15.0 | 22.9 | 13.2
  Week 8: A little worse: number analyzed (Participants) | 40 | 35 | 38
  Week 8: A little worse | 7.5 | 17.1 | 2.6
  Week 8: Much worse: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Much worse | 2.5 | 2.9 | 0
  Week 8: Very much worse: number analyzed (Participants) | 40 | 35 | 38
  Week 8: Very much worse | 5.0 | 0 | 0
  Week 12: Very much better: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Very much better | 5.9 | 2.9 | 5.6
  Week 12: Much better: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Much better | 20.6 | 22.9 | 25.0
  Week 12: A little better: number analyzed (Participants) | 34 | 35 | 36
  Week 12: A little better | 47.1 | 31.4 | 47.2
  Week 12: No change: number analyzed (Participants) | 34 | 35 | 36
  Week 12: No change | 14.7 | 17.1 | 16.7
  Week 12: A little worse: number analyzed (Participants) | 34 | 35 | 36
  Week 12: A little worse | 5.9 | 14.3 | 2.8
  Week 12: Much worse: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Much worse | 2.9 | 8.6 | 2.8
  Week 12: Very much worse: number analyzed (Participants) | 34 | 35 | 36
  Week 12: Very much worse | 2.9 | 2.9 | 0
  Week 20: Very much better: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Very much better | 2.9 | 11.4 | 10.5
  Week 20: Much better: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Much better | 28.6 | 17.1 | 34.2
  Week 20: A little better: number analyzed (Participants) | 35 | 35 | 38
  Week 20: A little better | 40.0 | 40.0 | 28.9
  Week 20: No change: number analyzed (Participants) | 35 | 35 | 38
  Week 20: No change | 20.0 | 20.0 | 15.8
  Week 20: A little worse: number analyzed (Participants) | 35 | 35 | 38
  Week 20: A little worse | 8.6 | 8.6 | 10.5
  Week 20: Much worse: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Much worse | 0 | 0 | 0
  Week 20: Very much worse: number analyzed (Participants) | 35 | 35 | 38
  Week 20: Very much worse | 0 | 2.9 | 0
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.8338, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = 0.01, 90% CI 2-sided [-0.19 to 0.20] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.1142, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.12, 90% CI 2-sided [-0.31 to 0.09] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.3433, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.20, 90% CI 2-sided [-0.38 to 0.00] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.1129, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.17, 90% CI 2-sided [-0.37 to 0.04] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.2842, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.20, 90% CI 2-sided [-0.38 to 0.00] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.0212, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.34, 90% CI 2-sided [-0.52 to -0.13] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.7665, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.07, 90% CI 2-sided [-0.28 to 0.14] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.1777, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.22, 90% CI 2-sided [-0.42 to -0.00] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.3741, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.12, 90% CI 2-sided [-0.33 to 0.09] — Somers'D statistic and tanh^(-1) transformed 90% CI
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.3321, Cochran-Mantel-Haenszel — Adjusted P-value obtained from Cochran-Mantel-Haenszel test (ANOVA for row means), adjusting for facial IGA at baseline; Risk Difference (RD) = -0.13, 90% CI 2-sided [-0.33 to 0.09] — Somers'D statistic and tanh^(-1) transformed 90% CI

12. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index Questionnaire (DLQI) Total Score at Weeks 2, 4, 8, 12, and 20
Description: DLQI was a simple 10-question validated questionnaire, each question was scored from 0 (not relevant/not at all) to 3 (very much). The DLQI total score ranged from 0 (no effect on participant's life) to 30 (extremely large effect on participant's life). The aim of this participant-reported questionnaire was to measure how much the skin condition had affected the participant's quality of life. The DLQI was administered to participants ≥ 16 years of age. Participants were administered the same questionnaire during the entire study based on their age at Day 1.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 27 | 26 | 24
units on a scale
  Change at Week 2 | -1.6 (4.53) | -1.9 (5.28) | -2.0 (3.37)
  Change at Week 4: number analyzed (Participants) | 25 | 25 | 24
  Change at Week 4 | -2.6 (5.01) | -3.6 (5.20) | -2.3 (4.19)
  Change at Week 8: number analyzed (Participants) | 27 | 25 | 24
  Change at Week 8 | -3.4 (5.28) | -4.0 (6.26) | -4.3 (4.93)
  Change at Week 12: number analyzed (Participants) | 21 | 24 | 23
  Change at Week 12 | -4.2 (4.71) | -2.9 (5.14) | -4.0 (4.98)
  Change at Week 20: number analyzed (Participants) | 22 | 26 | 24
  Change at Week 20 | -1.8 (5.75) | -3.7 (4.11) | -4.7 (5.69)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.7932, LRMM — LS Mean, SE, 90% CI, & p-value was based on a LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline DLQI as continuous covariate; LS Mean Difference = 0.3, 90% CI 2-sided [-1.56 to 2.14], Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.4365, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 0.9, 90% CI 2-sided [-0.99 to 2.73], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.8543, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = -0.2, 90% CI 2-sided [-1.92 to 1.54], Standard Error of Mean 1.04
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.8726, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = -0.2, 90% CI 2-sided [-1.91 to 1.58], Standard Error of Mean 1.05
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.5983, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 0.6, 90% CI 2-sided [-1.22 to 2.35], Standard Error of Mean 1.07
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.3396, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 1.0, 90% CI 2-sided [-0.77 to 2.86], Standard Error of Mean 1.09
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.5305, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = -0.6, 90% CI 2-sided [-2.23 to 1.01], Standard Error of Mean 0.97
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.0819, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 1.7, 90% CI 2-sided [0.09 to 3.29], Standard Error of Mean 0.96
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.0243, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 2.5, 90% CI 2-sided [0.69 to 4.31], Standard Error of Mean 1.09
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.1061, LRMM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 1.7, 90% CI 2-sided [-0.03 to 3.46], Standard Error of Mean 1.05

13. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Total Score at Weeks 2, 4, 8, 12, and 20
Description: CDLQI was a simple 10-question validated questionnaire, each question was scored from 0 (not relevant/not at all) to 3 (very much). The CDLQI total score ranged from 0 (no effect on participant's life) to 30 (extremely large effect on participant's life). The aim of this participant-reported questionnaire was to measure how much the skin condition had affected the participant's quality of life. The CDLQI was administered to participants < 16 years of age. Participants were administered the same questionnaire during the entire study based on their age at Day 1.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 14
units on a scale
  Change at Week 2: number analyzed (Participants) | 12 | 12 | 13
  Change at Week 2 | -1.6 (3.70) | -0.7 (9.00) | -2.0 (5.07)
  Change at Week 4 | -0.3 (2.90) | -2.7 (6.31) | -2.6 (4.69)
  Change at Week 8: number analyzed (Participants) | 12 | 9 | 14
  Change at Week 8 | -1.8 (4.52) | -2.2 (6.48) | -2.9 (4.85)
  Change at Week 12: number analyzed (Participants) | 12 | 10 | 13
  Change at Week 12 | -2.3 (4.46) | -1.1 (7.20) | -3.2 (4.67)
  Change at Week 20: number analyzed (Participants) | 11 | 8 | 14
  Change at Week 20 | -3.1 (4.44) | -3.5 (7.33) | -2.8 (4.71)
Statistical Analysis 1: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 2; Test type: Superiority; p = 0.9333, LRMM — LS Mean, SE, 90% CI, & p-value was based on a LRMM which included treatment, visit, treatment by visit interaction & facial IGA at baseline (Grade 3 vs. 4) as categorical covariates & baseline CDLQI as continuous covariate; LS Mean Difference = 0.1, 90% CI 2-sided [-2.69 to 2.97], Standard Error of Mean 1.67
Statistical Analysis 2: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 2; Test type: Superiority; p = 0.3972, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.4, 90% CI 2-sided [-1.40 to 4.27], Standard Error of Mean 1.67
Statistical Analysis 3: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 4; Test type: Superiority; p = 0.0662, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.1, 90% CI 2-sided [0.23 to 3.99], Standard Error of Mean 1.11
Statistical Analysis 4: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 4; Test type: Superiority; p = 0.8898, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.2, 90% CI 2-sided [-1.73 to 2.04], Standard Error of Mean 1.11
Statistical Analysis 5: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 8; Test type: Superiority; p = 0.3664, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.0, 90% CI 2-sided [-0.85 to 2.82], Standard Error of Mean 1.06
Statistical Analysis 6: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 8; Test type: Superiority; p = 0.0655, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.1, 90% CI 2-sided [0.25 to 4.05], Standard Error of Mean 1.10
Statistical Analysis 7: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 12; Test type: Superiority; p = 0.6921, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.5, 90% CI 2-sided [-1.61 to 2.57], Standard Error of Mean 1.20
Statistical Analysis 8: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 12; Test type: Superiority; p = 0.0406, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.7, 90% CI 2-sided [0.59 to 4.88], Standard Error of Mean 1.23
Statistical Analysis 9: Comparison: Imsidolimab 400/200 mg vs Placebo; Imsidolimab 400/200 mg vs Placebo: Week 20; Test type: Superiority; p = 0.6872, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.4, 90% CI 2-sided [-2.24 to 1.38], Standard Error of Mean 1.04
Statistical Analysis 10: Comparison: Imsidolimab 200/100 mg vs Placebo; Imsidolimab 200/100 mg vs Placebo: Week 20; Test type: Superiority; p = 0.3392, LRMM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.1, 90% CI 2-sided [-0.81 to 2.92], Standard Error of Mean 1.08

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment that did not necessarily have a causal relationship with treatment. An AE was considered "serious" if it resulted in death, life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, other important medical events. TEAE was defined as a new event that occurred during or after first dose of study treatment or any event present at baseline that worsens in either intensity or frequency after first dose of study treatment.
Time Frame: First dose of study drug until end of study (up to 20 weeks)
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Number analyzed (Participants) | 41 | 39 | 41
participants
  Any TEAEs | 18 | 10 | 11
  Serious TEAEs | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Randomization until end of study (up to 20 weeks) Adverse events: From first dose of study drug until end of study (up to 20 weeks)
Description: All-cause mortality: ITT Analysis Set
  Adverse events: Safety Analysis Set
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 8/41 | 6/39 | 6/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imsidolimab 400/200 mg (N=41) | Imsidolimab 200/100 mg (N=39) | Placebo (N=41)
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imsidolimab 400/200 mg (N=41) | Imsidolimab 200/100 mg (N=39) | Placebo (N=41)
COVID-19 (Infections and infestations) | 3 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 1
Headache (Nervous system disorders) | 3 | 0 | 0
Migraine (Nervous system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04856917/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04856917/SAP_001.pdf